CLINICAL TRIAL: NCT06754293
Title: Evaluating the Efficacy of Structured Exercise Interventions in Alleviating Aromatase Inhibitor-Induced Arthralgia in Breast Cancer Survivors: a Pilot Study Protocol
Acronym: RE-MS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Collaborators: Shanghai Cancer Hospital, China (Other)
Responsible Party: Principal Investigator, Lingyun Jiang, Principal Investigator, Fudan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 138103810480184013133114411411
Record Dates: First submitted 2024-11-24; First posted 2024-12-31 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-11

CONDITIONS: Musculoskeletal Symptoms; Breast Cancer; Endocrine Therapy; Aromatase Inhibitors
MeSH Terms: conditions — Breast Neoplasms | interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessors will be blinded to participant group assignments to ensure unbiased evaluation of study endpoints. Group allocation will be securely randomized, with access restricted to personnel uninvolved in assessments. Assessors will interact with participants following standardized protocols and receive de-identified data to prevent unintentional unmasking. Study staff will be trained to avoid disclosing treatment allocation during interactions. Any breach of masking will be documented, and corrective actions, such as reassignment or bias evaluation, will be implemented to maintain data integrity.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercise group (Experimental): The intervention group will participate in a home-based exercise program alongside standard rehabilitation guidance. Patients will receive exercise materials developed by the intervention team, along with a detailed explanation of the program, including its components, specific exercises, and expected benefits.The exercise program focuses on aerobic warm-ups and functional training, targeting key areas such as the hands, arms, shoulders, hips, legs, and back. It is designed to meet the rehabilitation needs of breast cancer patients undergoing endocrine therapy after surgery, addressing their unique challenges and enhancing recovery.The intervention team, composed of specialists in breast cancer treatment, rehabilitation therapists, nursing experts, and methodologists, has created a professional exercise guidance manual. This manual provides detailed descriptions of exercise types, specific methods, and safety precautions. To ensure effective implementation, instructional videos ha
  Interventions: Behavioral: rehabilitation exercise
- control group (No Intervention): Patients in the control group will receive standard guidance related to breast cancer endocrine therapy, including general information on exercise rehabilitation for managing bone and joint symptoms. This guidance allows patients the flexibility to choose their preferred form, type, and intensity of exercise. In addition, psychological counseling and health education will be provided to support their overall well-being.
  Monthly telephone follow-ups will be conducted to address concerns regarding the side effects of endocrine therapy. However, no specific exercise plans will be offered, nor will there be any monitoring or supervision of patients' adherence to exercise routines.

INTERVENTIONS:
Behavioral: rehabilitation exercise — The intervention group will participate in a home-based exercise program alongside standard rehabilitation guidance. Patients will receive exercise materials developed by the intervention team, along with a detailed explanation of the program, including its components, specific exercises, and expected benefits.
  The exercise program focuses on aerobic warm-ups and functional training, targeting key areas such as the hands, arms, shoulders, hips, legs, and back. It is designed to meet the rehabilitation needs of breast cancer patients undergoing endocrine therapy after surgery, addressing their unique challenges and enhancing recovery.
  The intervention team, composed of specialists in breast cancer treatment, rehabilitation therapists, nursing experts, and methodologists, has created a professional exercise guidance manual. This manual provides detailed descriptions of exercise types, specific methods, and safety precautions. To ensure effective implementation, instructional videos have
  Other Names: health education
  Arms: Exercise group

SUMMARY:
Endocrine therapy represents a foundational approach for managing hormone receptor-positive breast cancer, with treatment typically spanning 5 to 10 years. Although its clinical efficacy is well-established, medications like aromatase inhibitors frequently result in musculoskeletal (MS) complications, such as joint discomfort, stiffness (especially in the morning), carpal tunnel syndrome, tenosynovitis, myalgia, and reduced muscle strength. These issues, which can manifest intermittently or persistently, impact both central joints (spine, hips, shoulders) and peripheral ones (elbows, wrists, knees, feet), thereby substantially diminishing patients' quality of life (QoL). Evidence suggests that physical activity can mitigate these symptoms; however, adherence to exercise routines remains insufficient. Moreover, there is no agreement regarding the most effective type, intensity, or duration of exercise, and standardized guidelines are absent. Acknowledging the need for exercise as a sustainable habit, this research aims to design a home-based rehabilitation program customized for individuals undergoing endocrine therapy.

ELIGIBILITY:
Inclusion Criteria:1. Pathologically confirmed hormone receptor-positive breast cancer (stage I, II, III).

2. Initiation of treatment with aromatase inhibitors (e.g., anastrozole, letrozole, exemestane).

3. Postmenopausal women, including those with surgically induced menopause. 4. Clear consciousness, no cognitive or communication impairments, and able to comply with the intervention.

5. Informed consent obtained, with voluntary participation in the study. 6. Bone and joint symptoms with a Brief Pain Inventory (BPI) score of ≥3, or presence of at least one of the following risk factors: elevated bone turnover markers, reduced vitamin D levels, increased inflammatory cytokines, elevated C-reactive protein, or elevated rheumatoid factor.

7. Not participating in any physical therapy or exercise-based interventions that may interfere with this study.

-

Exclusion Criteria:

- 1. Recurrence of breast cancer or distant metastasis. 2. Presence of other malignancies. 3. Diagnosed rheumatoid arthritis, bone and joint trauma, or other severe bone and joint diseases.

4. Bone mineral density T-score <-2.5. 5. Presence of absolute contraindications to exercise.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
WOMAC | Baseline and 1month
  Developed in 1988 by Bellamy and Buchanan, the WOMAC index evaluates pain, stiffness, and physical function in knee or hip osteoarthritis patients over the past 48 hours . The WOMAC 3.1 version contains 24 items scored using either a VAS (0-100 mm) or a 5-point Likert scale (0-4). This study will use the VAS version, with pain (5 items, 0-500 points), stiffness (2 items, 0-200 points), and physical function (17 items, 0-1700 points) subscales. Total scores range from 0 to 2400, with higher scores indicating greater symptom burden. Scores below 800 denote mild symptoms, 800-1200 moderate, and above 1200 severe symptoms.
Grip strength | Baseline and 1month
  Grip strength will be measured by the exercise group at baseline (0 months) and at 1, 3, and 6 months of intervention. An electronic hand dynamometer (CAMRY EH10) will be used for assessment. Participants will perform the test by extending their arms straight down with their palms facing their thighs, abducting their dominant upper limb (on the non-surgical side) by 30 degrees. The grip strength value, displayed in kilograms on the dynamometer, will represent the maximum force achieved. To ensure accuracy, participants will be instructed not to swing their arms, squat, or allow the dynamometer to touch their body during the test. Each participant will undergo three assessments, with a 60-second interval between measurements, and the highest value will be used for analysis.
M-SACRAH | Baseline and 1month
  The SACRAH, developed by Leeb et al. in 2003, is a validated tool for assessing chronic rheumatic hand conditions. The Modified Score for the Assessment of Chronic Rheumatoid Affections of the Hands (M-SACRAH), a shorter and simplified version of SACRAH, has shown similar reliability and representativeness. M-SACRAH contains 12 items scored using a visual analog scale (VAS, 0-100 mm) across three dimensions: pain (2 items, 0-200 points), stiffness (2 items, 0-200 points), and physical function (8 items, 0-800 points). Higher scores indicate more severe symptoms, with a total possible score of 0-1200.
BCTQ | Baseline and 1month
  The BCTQ consists of 11 items assessing symptom severity (Symptom Severity Score, SSS) and 8 items evaluating functional status (Function Scale Score, FSS) . The SSS addresses issues such as nocturnal pain, frequency of night awakenings, daytime wrist pain, hand numbness or weakness, and difficulty handling small objects. The FSS evaluates activities like writing, buttoning clothes, carrying groceries, and performing household tasks. Each item is rated on a 5-point scale, with 1 indicating "none" and 5 indicating "severe." The average score across all items represents the final score.
Range of Motion | Baseline and 1month
  Tools for ROM measurement include goniometers, rulers, and electronic measuring devices. The goniometer comprises a stationary arm (proximal arm) with a semicircular (0°-180°) or circular (0°-360°) angle scale and a movable arm (distal arm) attached via a rivet. The movable arm rotates with the limb, allowing ROM to be read from the scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Cancer Center, Shanghai, XuHui, China

IPD SHARING:
Plan to Share IPD: No